CLINICAL TRIAL: NCT01947335
Title: Minimizing cOntrast utiliZAtion With IVUS Guidance in coRonary angioplasTy: The MOZART Study
Brief Title: IVUS Guidance to Reduce Contrast in Coronary Angioplasty
Acronym: MOZART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Pedro A. Lemos, Professor of Medicine, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02358512.7.0000.0068
Record Dates: First submitted 2013-01-01; First posted 2013-09-20 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-05

CONDITIONS: Contrast Media Reaction; Acute Renal Failure
Keywords: Coronary; Angioplasty; Percutaneous coronary intervention; Stent; Contrast; Acute Renal failure; Intravascular ultrasound; Prevention
MeSH Terms: conditions — Acute Kidney Injury | interventions — Ultrasonography, Interventional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Angiography-guided PCI (No Intervention): Angiography-guided percutaneous coronary intervention
- IVUS-guided PCI (Active Comparator): Intravascular ultrasound guided percutaneous coronary intervention
  Interventions: Device: IVUS-guided PCI

INTERVENTIONS:
Device: IVUS-guided PCI — Intravascular ultrasound guided percutaneous coronary intervention
  Other Names: Intravascular ultrasound
  Arms: IVUS-guided PCI

SUMMARY:
This study tests the hypothesis that ultrasound-guided PCI reduces contrast volume during the procedure.

DETAILED DESCRIPTION:
Contrast-induced acute kidney injury (CI-AKI) is an important adverse effect of percutaneous coronary interventions. Despite various efforts, very few preventive measures have been shown effective in reducing its incidence. The final volume of contrast media utilized during the procedure is a well-known independent factor affecting the occurrence of CI-AKI.

Intravascular ultrasound (IVUS) has been largely used as an adjunctive diagnostic tool during percutaneous coronary intervention (PCI). When fully explored, IVUS provides precise information for guiding the PCI strategy. IVUS allows accurate vessel and lesion sizing, determination of plaque calcification (and the need for pre-stent plaque preparation), assessment of post-stent results (including edge dissections and residual lesion, as well as stent underexpansion or incomplete apposition). Therefore, IVUS has the potential to reduce the utilization of contrast media during PCI.

In the present study, we hypothesize that IVUS guidance is associated with a significant reduction in the volume of contrast media during PCI, in comparison to standard angiography-guided intervention.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age >=18 years
* Coronary artery disease scheduled for percutaneous intervention
* Technical feasibility for intravascular ultrasound to guide coronary angioplasty
* Increased risk for contrast-induced acute renal failure (e.g. age > 80 years, female gender, diabetes, urgent or emergent procedure priority, diabetes, congestive heart failure, increased baseline serum creatinine, decreased calculated or measured creatinine clearance, intra-aortic balloon pumping, previous renal transplantation or single kidney)

Exclusion Criteria:

* Anticipated technical impossibility for intravascular ultrasound
* Unknown baseline renal function
* Baseline end-stage renal failure needing dialysis
* Acute renal failure with dynamic change in renal function at the time of index procedure
* Iodine contrast administration <= 72 prior to index procedure
* Known allergy to iodine contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro A Lemos, MD PhD, Study Chair — Heart Institute - InCor. University of Sao Paulo Medical School; Paulo R Soares, MD PhD, Principal Investigator — Heart Institute - InCor. University of Sao Paulo Medical School
Locations (1):
- Heart Institute - InCor. University of Sao Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Mariani J Jr, Guedes C, Soares P, Zalc S, Campos CM, Lopes AC, Spadaro AG, Perin MA, Filho AE, Takimura CK, Ribeiro E, Kalil-Filho R, Edelman ER, Serruys PW, Lemos PA. Intravascular ultrasound guidance to minimize the use of iodine contrast in percutaneous coronary intervention: the MOZART (Minimizing cOntrast utiliZation With IVUS Guidance in coRonary angioplasTy) randomized controlled trial. JACC Cardiovasc Interv. 2014 Nov;7(11):1287-93. doi: 10.1016/j.jcin.2014.05.024. Epub 2014 Oct 15. PMID 25326742

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Angiography-guided PCI | IVUS-guided PCI
Started | 42 | 41
Completed | 42 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Angiography-guided PCI | IVUS-guided PCI | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Continuous [Median (Full Range); unit: years] | 62.1 [57.3 to 76.5] | 67.1 [58.3 to 76.1] | 64.6 [57.3 to 76.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 24 | 24 | 48
Region of Enrollment [Number; unit: participants]
  Brazil | 42 | 41 | 83

OUTCOME MEASURES:

1. Primary Outcome: Total Volume of Iodine Contrast Used During Procedure
Description: Total volume of iodine contrast administered during the index procedure.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Angiography-guided PCI | IVUS-guided PCI
Number analyzed (Participants) | 42 | 41
ml | 64.5 [42.8 to 97.0] | 20.0 [12.5 to 30]

2. Secondary Outcome: Major Adverse Cardiac Events
Description: Composite of death, myocardial infarction or repeat revascularization
Time Frame: 30 days and 6 months
Measure: Number; unit: participants
Arm/Group | Angiography-guided PCI | IVUS-guided PCI
Number analyzed (Participants) | 42 | 41
participants
  30 days | 2 | 2
  6-months | 2 | 5

3. Secondary Outcome: Incidence of Contrast-induced Nephropathy
Description: Increase >= 0.5 mg/dl in basal serum creatinine
Time Frame: 7 days
Measure: Number; unit: percentage of participants
Arm/Group | Angiography-guided PCI | IVUS-guided PCI
Number analyzed (Participants) | 42 | 41
percentage of participants | 19 | 7.3

ADVERSE EVENTS:
Time Frame: In-hospital
Arm/Group | Angiography-guided PCI | IVUS-guided PCI
Serious Adverse Events (participants affected / at risk) | 2/42 | 2/41
Other Adverse Events (participants affected / at risk) | 8/42 | 3/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Angiography-guided PCI (N=42) | IVUS-guided PCI (N=41)
Periprocedural Infarction (Cardiac disorders) | 2 (2) | 2 (2)
Unplanned revascularization (Cardiac disorders) | 0 (0) | 0 (0)
Stent Thrombosis (Cardiac disorders) | 0 (0) | 0 (0)
Death (Cardiac disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Angiography-guided PCI (N=42) | IVUS-guided PCI (N=41)
Peak increase in creatinine > 0.5mg/dl (Renal and urinary disorders) | 8 (8) | 3 (3) — Peak increase in creatinine > 0.5mg/dl

LIMITATIONS AND CAVEATS:
Patients were enrolled according to somewhat restricted criteria, which excluded patients with recent catheterization, using nephrotoxic agents, or with unstable or unknown renal function.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No